CLINICAL TRIAL: NCT04833400
Title: Intelligent Cardiopulmonary Rehabilitation System for Patients With Chronic Stroke: a Feasibility Study
Brief Title: Intelligent Cardiopulmonary Rehabilitation System for Patients With Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Physical Medicine and Rehabilitation, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N202010012
Record Dates: First submitted 2021-01-03; First posted 2021-04-06 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Stroke
Keywords: cardiopulmonary exercise; cardiorespiratory fitness; aerobic training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intelligent cardiopulmonary rehabilitation system (ICRS) (Experimental): The ICRS is very likely to the conventional stationary biking, but with an algorithm that automatically controls the resistance of pedalling, considering the instant heart rate and cadence, to keep the heart rate within the targeted heart rate zone.
  Interventions: Device: ICRS
- Traditional aerobic exercise training (TAET) (Active Comparator): The TAET is performed with stationary biking, with intensity being set as subjective rating of perceived exertion at a "somewhat hard" to "hard" level. The resistance of pedaling is ad-justed by the user or physical therapist.
  Interventions: Device: TAET

INTERVENTIONS:
Device: ICRS — Patients undergo 30-minute aerobic training with ICRS, 3 sessions a week, for 4 weeks.
  Arms: Intelligent cardiopulmonary rehabilitation system (ICRS)
Device: TAET — Patients undergo 30-minute aerobic training with TAET, 3 sessions a week, for 4 weeks.
  Arms: Traditional aerobic exercise training (TAET)

SUMMARY:
By comparing with traditional aerobic exercise training (TAET), we investigate the effects of an intelligent cardiopulmonary rehabilitative system (ICRS) on cardiopulmonary fitness and patient satification among patients with chronic stroke.

DETAILED DESCRIPTION:
Cycle ergometer training is one of the common indoor aerobic exercises for enhancing cardiorespiratory fitness in patients after stroke. However, studies had suggested that patients may be undertrained for reasons such as a tight time schedule for other rehabilitation programs and lack of objective evaluation on the training intensity.

To address the issue of inadequate cycle ergometer training in poststroke patients, in this study, an intelligent cardiopulmonary rehabilitation system was developed and incorporated into a bicycle ergometer, allowing dynamically auto-adjust paddling resistance considering the instant heart rate and cadence, with a goal to maintain the hear rate within the pre-determined heart rate zone. The purpose of the current study is to investigate the feasibility of the ICRS in stroke patients and whether it outweighs the traditional feedback on training intensity.

A single-blind crossover trial is adopted with 40 participants estimated to be recruited and randomly assigned to the group A and group B. Group A received training with ICRS while Group B received training with TAET at the beginning. The intensity of ICRS is set as 60%~80% heart rate reserve (HRR) which is obtained from cardiopulmonary exercise testing (CPET) at pretest. The intensity of TAET is set as subjective rating of perceived exertion at "somewhat hard" to "hard" level. Both groups will receive 30 minutes of training per session, 3 sessions a week for four weeks followed by a washout period of 4-week break. Subjects are crossed-over to the alternate treatment afterwards. CPET evaluations will be conducted in a total of 4 times before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-75 y/o
* Healthy people
* Chronic stroke > 6 months
* Able to walk independently > 6 minutes with or without orthosis
* Able to use stationary bike
* MRS(Modified Rankin Scale) ranged 1 to 3

Exclusion Criteria:

* Patients whose heart rate can not be used as the indicator of training intensity (eg, ar-rhythmia, atrial fibrillation, beta-blockers users)
* With any reason that the patient is not suitable to undergo aerobic training
* Patients who are unable to do cycling due to musculoskeletal problems
* Patients who can not follow the instruction of trainers due to cognitive or emotional-problems.
* Patients whose medical condition is not unstable.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
relative VO2-peak (mL/kg/min) | 4 weeks
  oxygen consumption (VO2- peak) is measured during a the cardiopulmonary exercise test with a ramped stationary biking.

SECONDARY OUTCOMES:
6-min walk test | 4 weeks
  The 6-minute walk test measures the distance covered while walking at a tolerable pace for 6 minutes.
absolute VO2-peak (mL/min) | 4 weeks
  oxygen consumption (VO2- peak) is measured during a the cardiopulmonary exercise test with a ramped stationary biking.
workload-peak (Watt) | 4 weeks
  The peak workload is measured during a the cardiopulmonary exercise test with a ramped stationary biking.

CONTACTS AND LOCATIONS:
Locations (1):
- WanFang Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No